CLINICAL TRIAL: NCT00432237
Title: A Phase III, Multicenter, Randomized, Placebo-Controlled Clinical Trial to Study the Safety and Efficacy of Oral MK0974 in the Acute Treatment of Migraine With or Without Aura
Brief Title: Safety and Efficacy Study of MK0974 in the Acute Migraine (0974-016)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0974-016; 2006_526
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Results first posted 2010-12-06 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — telcagepant

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- MK0974 50 mg (Experimental): MK0974 50 mg; one orally-administered dose, plus an optional second dose (MK0974 50 mg) to treat a single moderate-to-severe migraine attack
  Interventions: Drug: MK0974 50 mg
- MK0974 150 mg (Experimental): MK0974 150 mg; one orally-administered dose, plus an optional second dose (MK0974 150 mg) to treat a single moderate-to-severe migraine attack
  Interventions: Drug: MK0974 150 mg
- MK0974 300 mg (Experimental): MK0974 300 mg; one orally-administered dose, plus an optional second dose (MK0974 300 mg or placebo) to treat a single moderate-to-severe migraine attack
  Interventions: Drug: MK0974 300 mg
- Placebo (Placebo Comparator): Placebo; one orally-administered dose, plus an optional second dose (placebo) to treat a single moderate-to-severe migraine attack
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK0974 50 mg
  Other Names: MK0974
  Arms: MK0974 50 mg
Drug: MK0974 150 mg
  Other Names: MK0974
  Arms: MK0974 150 mg
Drug: MK0974 300 mg
  Other Names: MK0974
  Arms: MK0974 300 mg
Drug: Comparator: Placebo — MK0974 50 mg soft gel capsule Placebo; MK0974 150 mg soft gel capsule Placebo; MK0974 300 mg soft gel capsule Placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of MK0974 compared to a placebo for acute migraine.

ELIGIBILITY:
Inclusion Criteria:

* Patient has at least 1 year history of migraine (with or without aura)
* Females of childbearing years must use acceptable contraception throughout trial

Exclusion Criteria:

* Patient is pregnant/breast-feeding (or is a female expecting to conceive during the study period)
* Patient has history or evidence of uncontrolled diabetes, or Human Immunodeficiency Virus (HIV) disease. Patient has uncontrolled cardiovascular disease
* Patient has major depression, other pain syndromes that might interfere with study assessments, psychiatric conditions, dementia, or significant neurological disorders (other than migraine)
* Patient has a history of gastric or small intestinal surgery or has a disease that causes malabsorption
* Patient has a history of cancer within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1703 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Connor KM, Shapiro RE, Diener HC, Lucas S, Kost J, Fan X, Fei K, Assaid C, Lines C, Ho TW. Randomized, controlled trial of telcagepant for the acute treatment of migraine. Neurology. 2009 Sep 22;73(12):970-7. doi: 10.1212/WNL.0b013e3181b87942. PMID 19770473

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 83 centers worldwide that participated: United States (36), Latin America (9), and Europe (38). First Patient Treated = 25 March 2007, and Last Patient Last Treatment = 29 November 2007.
Pre-assignment Details: Participants were assessed, using the protocol inclusion and exclusion criteria, at Visit 1, and if eligible were randomized at that same visit.
Period: Overall Study
Arm/Group | MK0974 50 mg | MK0974 150 mg | MK0974 300 mg | Placebo
Started | 244 (1 patient in the MK0974 50 mg group was treated but withdrew consent.) | 485 | 484 (1 patient in the MK0974 300 mg group was treated but withdrew consent.) | 490
Completed--With Data | 176 | 381 | 370 | 365
Completed--No Data | 1 (For patients in this category, diaries were collected but lost prior to data entry.) | 3 (For patients in this category, diaries were collected but lost prior to data entry.) | 5 (For patients in this category, diaries were collected but lost prior to data entry.) | 1 (For patients in this category, diaries were collected but lost prior to data entry.)
Completed | 177 | 384 | 375 | 366
Not Completed | 67 | 101 | 109 | 124
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 10 | 10 | 18 | 18
Not completed — Physician Decision | 1 | 3 | 2 | 1
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 13 | 10 | 11 | 8
Not completed — Withdrawal by Subject | 5 | 6 | 9 | 11
Not completed — Lack of Qualifying Event | 38 | 71 | 69 | 84

BASELINE CHARACTERISTICS:
Groups:
- MK0974 50 mg: MK0974 50 mg; one orally-administered dose, plus an optional second dose (MK0974 50 mg) to treat a single moderate-to-severe migraine attack
  The reported number of participants are all patients randomized who received study drug and completed the study.
- MK0974 150 mg: MK0974 150 mg; one orally-administered dose, plus an optional second dose (MK0974 150 mg) to treat a single moderate-to-severe migraine attack
  The reported number of participants are all patients randomized who received study drug and completed the study.
- MK0974 300 mg: MK0974 300 mg; one orally-administered dose, plus an optional second dose (MK0974 300 mg or placebo) to treat a single moderate-to-severe migraine attack
  The reported number of participants are all patients randomized who received study drug and completed the study.
- Placebo: Placebo; one orally-administered dose, plus an optional second dose (placebo) to treat a single moderate-to-severe migraine attack
  The reported number of participants are all patients randomized who received study drug and completed the study.
- Total: Total of all reporting groups
Arm/Group | MK0974 50 mg | MK0974 150 mg | MK0974 300 mg | Placebo | Total
Number analyzed (Participants) | 177 | 381 | 371 | 365 | 1294
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline Characteristics are for the subset of randomized patients who were treated
  years | 41.4 (11.3) | 41.6 (11.0) | 41.8 (11.6) | 41.9 (11.9) | 41.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline Characteristics are for the subset of randomized patients who were treated
  Participants
    Female | 156 | 329 | 320 | 318 | 1123
    Male | 21 | 52 | 51 | 47 | 171
Race/Ethnicity, Customized [Number; unit: participants] — Baseline Characteristics are for the subset of randomized patients who were treated
  participants
    White | 148 | 320 | 302 | 303 | 1073
    Black | 10 | 16 | 23 | 20 | 69
    Asian | 1 | 6 | 1 | 8 | 16
    American Indian or Alaska Native | 1 | 2 | 0 | 0 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
    Multi-Racial | 17 | 37 | 44 | 33 | 131
    Missing | 0 | 0 | 0 | 1 | 1
Baseline Severity [Number; unit: Participants] — Baseline severity was self-reported by the patient and recorded in the take-home diary. Patients were instructed not to dose until they had experienced either a moderate or severe migraine, with migraine pain rated on a 4-point scale (No Pain=0, Mild Pain=1, Moderate Pain=2, Severe Pain=3). Baseline Characteristics are for the subset of randomized patients who were treated.
  Participants
    Moderate | 108 | 254 | 237 | 235 | 834
    Severe | 69 | 127 | 133 | 130 | 459
    Baseline Severity missing | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reporting Pain Freedom at 2 Hours Postdose
Description: Pain Freedom was defined as a reduction of a Grade 2 or 3 severity migraine at baseline to a no pain (Grade 0) at 2 hours post dose.
  Headache severity was recorded by the patient in a diary. 0=no pain; 1=mild pain; 2=moderate pain; 3=severe pain.
Time Frame: 2 hours post dose
Population: All randomized, treated patients who have at least one post-dose measurement at or prior to 2 hours.
Measure: Number; unit: Participants
Arm/Group | MK0974 50 mg | MK0974 150 mg | MK0974 300 mg | Placebo
Number analyzed (Participants) | 176 | 380 | 369 | 365
Participants | 29 | 88 | 88 | 39
Statistical Analysis 1: Comparison: MK0974 150 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; P-value constructed using a logistic model adjusting for baseline severity (moderate, severe), region (US, ex-US), treatment and age (continuous)
Statistical Analysis 2: Comparison: MK0974 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Patients Who Have Sustained Pain-Freedom From 2 to 24 Hours Postdose
Description: Pain Freedom at 2 hours postdose, with no administration of any rescue medication and no occurrence thereafter of a mild/moderate/severe headache during the 24 hours after dosing with study medication.
Time Frame: 2 to 24 hours postdose
Population: All randomized, treated patients who have at least one post-dose measurement at or prior to 2 hours and who either 1) did not have pain freedom at any time between 2 and 24 hours postdose, 2) used rescue medication between 2 and 24 hours postdose or 3) answered the 24 hour recurrence question (a question that ascertains recurrence of migraine pain)
Measure: Number; unit: Participants
Arm/Group | MK0974 50 mg | MK0974 150 mg | MK0974 300 mg | Placebo
Number analyzed (Participants) | 177 | 378 | 365 | 363
Participants | 25 | 62 | 63 | 26
Statistical Analysis 1: Comparison: MK0974 150 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK0974 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Number of Patients Reporting Pain Relief at 2 Hours Post Dose
Description: Reduction of a Grade 2 or 3 severity migraine at baseline to mild or no pain (Grade 1 or 0) at 2 hours post dose.
  Headache severity was recorded by the patient in a diary. 0=no pain; 1=mild pain; 2=moderate pain; 3=severe pain.
Time Frame: 2 hours post dose
Population: All randomized, treated patients who have at least one post-dose measurement at or prior to 2 hours.
Measure: Number; unit: Participants
Arm/Group | MK0974 50 mg | MK0974 150 mg | MK0974 300 mg | Placebo
Number analyzed (Participants) | 176 | 380 | 369 | 365
Participants | 78 | 205 | 205 | 120
Statistical Analysis 1: Comparison: MK0974 150 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK0974 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]

4. Primary Outcome: Number of Patients Reporting Absence of Photophobia at 2 Hours Post Dose
Description: Respective experience (yes/no) of migraine-associated symptoms (including photophobia) was recorded by the patient in a diary.
Time Frame: 2 hours post dose
Population: All randomized, treated patients who have at least one post-dose measurement at or prior to 2 hours.
Measure: Number; unit: Participants
Arm/Group | MK0974 50 mg | MK0974 150 mg | MK0974 300 mg | Placebo
Number analyzed (Participants) | 176 | 380 | 369 | 365
Participants | 72 | 176 | 179 | 119
Statistical Analysis 1: Comparison: MK0974 150 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK0974 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]

5. Primary Outcome: Number of Patients Reporting Absence of Phonophobia at 2 Hours Post Dose
Description: Respective experience (yes/no) of migraine-associated symptoms (including phonophobia) was recorded by the patient in a diary.
Time Frame: 2 hours post dose
Population: All randomized, treated patients who have at least one post-dose measurement at or prior to 2 hours.
Measure: Number; unit: Participants
Arm/Group | MK0974 50 mg | MK0974 150 mg | MK0974 300 mg | Placebo
Number analyzed (Participants) | 176 | 380 | 369 | 365
Participants | 85 | 192 | 206 | 152
Statistical Analysis 1: Comparison: MK0974 150 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK0974 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]

6. Primary Outcome: Number of Patients Reporting Absence of Nausea at 2 Hours Post Dose
Description: Respective experience (yes/no) of migraine-associated symptoms (including nausea) was recorded by the patient in a diary.
Time Frame: 2 hours post dose
Population: All randomized, treated patients who have at least one post-dose measurement at or prior to 2 hours.
Measure: Number; unit: Participants
Arm/Group | MK0974 50 mg | MK0974 150 mg | MK0974 300 mg | Placebo
Number analyzed (Participants) | 176 | 380 | 369 | 365
Participants | 113 | 260 | 258 | 196
Statistical Analysis 1: Comparison: MK0974 150 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK0974 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Patients Who Have Total Migraine Freedom 2 to 24 Hours Postdose
Description: Pain Freedom and no migraine-associated symptoms at 2 hours postdose, with no administration of any rescue medication and no occurrence thereafter of a mild/moderate/severe headache or migraine-associated symptom during the 24 hours after dosing with study medication.
Time Frame: 2 to 24 hours postdose
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | MK0974 50 mg | MK0974 150 mg | MK0974 300 mg | Placebo
Number analyzed (Participants) | 177 | 378 | 365 | 363
Participants | 20 | 55 | 54 | 23
Statistical Analysis 1: Comparison: MK0974 150 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK0974 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: Number of Patients Who Have Total Migraine Freedom 2 Hours Postdose
Description: Pain Freedom and no migraine-associated symptoms at 2 hours postdose.
Time Frame: 2 hours postdose
Population: All randomized, treated patients who have at least one post-dose measurement at or prior to 2 hours.
Measure: Number; unit: Participants
Arm/Group | MK0974 50 mg | MK0974 150 mg | MK0974 300 mg | Placebo
Number analyzed (Participants) | 176 | 380 | 369 | 365
Participants | 24 | 78 | 78 | 36
Statistical Analysis 1: Comparison: MK0974 150 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK0974 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time that the patient was first treated with study therapy through 14 days following the last dose of study therapy.
Description: Subjective adverse experiences were recorded by the patient in a paper diary.
  Patients were counted in the treatment group for which they actually took study drug. One patient gave some of their study drug to another patient; resulting in the difference in 2 groups of 1 from what was reported in the Participant Flow "Completed--With Data".
Arm/Group | MK0974 50 mg | MK0974 150 mg | MK0974 300 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/177 | 1/381 | 0/370 | 1/366
Other Adverse Events (participants affected / at risk) | 45/177 | 69/381 | 94/370 | 77/366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0974 50 mg (N=177) | MK0974 150 mg (N=381) | MK0974 300 mg (N=370) | Placebo (N=366)
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK0974 50 mg (N=177) | MK0974 150 mg (N=381) | MK0974 300 mg (N=370) | Placebo (N=366)
Vertigo (Ear and labyrinth disorders) | 3 | 2 | 5 | 10
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 4 | 12 | 6
Dry Mouth (Gastrointestinal disorders) | 9 | 17 | 19 | 19
Nausea (Gastrointestinal disorders) | 14 | 13 | 19 | 20
Vomiting (Gastrointestinal disorders) | 6 | 3 | 6 | 10
Fatigue (General disorders) | 9 | 15 | 25 | 14
Dizziness (Nervous system disorders) | 13 | 9 | 20 | 12
Headache (Nervous system disorders) | 0 | 3 | 3 | 8
Paraesthesia (Nervous system disorders) | 3 | 5 | 8 | 9
Somnolence (Nervous system disorders) | 7 | 14 | 10 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.